CLINICAL TRIAL: NCT05585879
Title: Outpatient Colonoscopy: Demonstrating Effective Salvage of Inadequate Colonoscopies Utilizing the Pure-Vu EVS System
Brief Title: Demonstrating Effective Salvage of Inadequate Colonoscopies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Strategy changed
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL00052
Record Dates: First submitted 2022-09-23; First posted 2022-10-19 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Screening

STUDY DESIGN:
Intervention Model Description: Multicenter, Prospective, Consecutive Series, Pragmatic Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pure-Vu EVS (Other): Rate of incomplete colonoscopies due to inadequate preparation salvaged to adequate colonoscopies with the use of the Pure-Vu EVS System.
  Inadequate OCs defined as such if any of the following are met:
  * BBPS < 6 (Adequacy is defined as BBPS of 2 or greater in each segment)
  * Inability to identify > 5mm polyps The estimated rate of salvaged preparations will be calculated and presented with exact one-sided 95% confidence interval: Number of preps inadequate with SOC and adequate after Pure-VU EVS System / Number of preps inadequate with SOC.
  The lower bound will be compared to a 35% performance goal.
  Interventions: Device: Pure-Vu EVS

INTERVENTIONS:
Device: Pure-Vu EVS — Subjects will be enrolled until 115 inadequate bowel prep cases via SOC are accrued and subsequently treated with Pure-Vu EVS. Inadequate OCs defined as such if any of the following are met:
  * Boston Bowel Preparation Score (BBPS) < 6 (Adequacy is defined as BBPS of 2 or greater in each segment)
  * Inability to identify > 5mm polyps

SUMMARY:
The aim of this study is to demonstrate that the use of the Pure-Vu EVS System can salvage inadequately prepared optical colonoscopies (OCs) to adequate OCs.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the reduction of inadequate colonoscopies when Pure-Vu EVS System is used to salvage inadequately prepped colons as defined by the multi-society guidelines (USMSTF).

ELIGIBILITY:
Inclusion Criteria:

1. Eligible adults aged between 40-80
2. Elective outpatient colonoscopy by participating gastroenterologist

Exclusion Criteria:

1. Not competent to consent
2. Known or suspected bleeding disorders such as, but not limited to hemophilia and von Willebrand disease
3. History of colonic resection
4. Prior incomplete colonoscopy due to patient anatomy
5. Diverticulitis
6. Active Inflammatory bowel disease (Crohn's, Ulcerative Colitis, or Indeterminate)
7. Known or suspected colon stricture
8. Hereditary Colorectal Cancer Syndrome
9. Subject is pregnant or suspected pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Rate of incomplete colonoscopies | Day 0 (Procedure Day)
  Rate of incomplete colonoscopies due to inadequate preparation salvaged to adequate colonoscopies with the use of the Pure-Vu EVS System.
  Inadequate OCs defined as such if any of the following are met:
  * BBPS < 6 (Adequacy is defined as BBPS of 2 or greater in each segment)
  * Inability to identify > 5mm polyps The estimated rate of salvaged preparations will be calculated and presented with exact one-sided 95% confidence interval: Number of preps inadequate with SOC and adequate after Pure-VU EVS System / Number of preps inadequate with SOC.
  The lower bound will be compared to a 35% performance goal.

SECONDARY OUTCOMES:
Assessment of Screening | Day 0 (Procedure Day)
  The following secondary endpoint will be assessed:
  Number of polyps and adenomas: type, location, size, pathology and morphology
Assessment of Screening | Day 0 (Procedure Day)
  Boston Bowel Prep Score (BBPS) before and after Pure-Vu EVS use. Throughout the procedure, the study endoscopist will be requested to document the pre-cleansing BBPS and post- cleansing BBPS for each colon segment.
Procedural Outcome | Day 0 (Procedure Day)
  Sedation type The type of sedation will not be dictated by the study but will be documented.
Procedural Outcome | Day 0 (Procedure Day)
  Cecum Intubation Rate
Assessment screening | Day 0 (Procedure Day)
  Polyp Miss Rate (PMR)
Assessment screening | Day 0 (Procedure Day)
  Adenoma Detection Rate (ADR)
Assessment screening | Day 0 (Procedure Day)
  Adenoma Miss Rate (AMR)
Assessment screening | Day 0 (Procedure Day)
  Adenoma Per Colonoscopy (APC)
Assessment screening | Day 0 (Procedure Day)
  Adenomas Per Positive Patient (APP)
Assessment screening | Day 0 (Procedure Day)
  Sessile Serrated Adenoma Detection Rate
Assessment Screening | Day 0 (Procedure Day)
  Polyp Detection Rate (PDR)
Procedural Outcomes | Day 0 (Procedure Day)
  Procedure Time: Time to cecum and withdrawal time
Procedural Outcomes | Day 0 (Procedure Day)
  Intraprocedural tools The type of Intraprocedural tools will not be dictated by the study but will be documented.

OTHER OUTCOMES:
User Satisfaction | Day 0(Procedure Day)
  Clinician Satisfaction Questionnaire: Each clinician will complete a questionnaire for each completed Pure-Vu EVS procedure.
Comparison Rates | Day 0 (Procedure Day) - 1-14 day follow up
  Comparison of SAE rates between Pure-Vu subjects and the published serious complication rate of standard colonoscopy procedures (2.8%)
Economic Impact | Through study completion, an average of 1 year.
  Economic Impact: Impact will be calculated by utilizing both data generated as part of the study and data published on the costs associated with outpatient colonoscopies and subsequent findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pomeranz, Study Director — Motus GI Medical Technologies Ltd
Locations (1):
- NYU, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Information regarding the study and study data will be made available via publication on clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of the study.
Access Criteria: clinicaltrials.gov
URL: http://www.clinicaltrials.gov

REFERENCES:
- See also: More information about Pure-VU® EVS — https://www.motusgi.com/physicians-nurses/pure-vu-system/

DOCUMENTS (1):
  • Study Protocol (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT05585879/Prot_001.pdf